CLINICAL TRIAL: NCT03697369
Title: Glycemic Control and Treatment Satisfaction in Children With Type 1 Diabetes Using Insulin Pumps
Status: Completed | Type: Observational
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Collaborators: Wolfson Medical Center (Other Government); Sheba Medical Center (Other Government); Maccabi Healthcare Services, Israel (Other)
Responsible Party: Sponsor
Other Study IDs: 0073-15-ASF
Record Dates: First submitted 2018-07-16; First posted 2018-10-05 (Actual); Last update posted 2018-10-05 (Actual); Status verified 2018-10

CONDITIONS: T1DM

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Observation group: Individuals with T1D ages 0-20 years who switched management modality from MDI to pump as part of their clinical care and were followed up prospectively in the next 12 months.

SUMMARY:
Background: The use of insulin pumps in pediatric patients with type 1 diabetes(T1D) has expanded, with lack of data comparing between the different devices.

Objective: to compare prospectively glycemic control, technical difficulties and quality of life (QOL) between 3 pump devices during the first year of use .

Methods: a prospective observational trial, based on clinical data retrieved during 12 months of follow- up. Inclusion criteria included T1D patients, ages 1-18 years, who started pump therapy as part of their clinical care in 4 university affiliated medical centers. The devices fully reimbursed by national health insurance are: MiniMed™ 640G , MiniMed® Veo™, Animas® Vibe®, and Abbott Omnipod®. Comparison parameters included quality of life (QOL), frequency of technical difficulties, skin reactions, discontinuation rate, glycated hemoglobin (HBA1C), mean glucose, total daily insulin dose (TDD) , pump setting parameters and BMI.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of T1D recorded by a pediatric endocrinologist
* Attending periodic clinic visits, and starting pump mode of therapy between May 2015 and March 2017.

Exclusion Criteria:

• No restrictions on HbA1c value at study recruitment or on use of CGMS -

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population included all individuals with T1D ages 0-20 years who switched management modality from MDI to pump as part of their clinical care, and were managed by the pediatric diabetes teams from the AWeSoMe Study Group ( four pediatric diabetes multidisciplinary clinics in Israel; Assaf Harofeh Medical Center, E. Wolfson Medical Center, Edmond and Lily Safra Children's Hospital, and Maccabi National Juvenile Diabetes Center).
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2015-05-31 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Technical difficulties differences | 2 years from patient first enrollment
  All patients were asked 5 questions regarding monthly frequency of technical problems including the need to use extra sets and the level of pain at catheter insertion
Quality Of Life (QOL) | 2 years from patient first enrollment
  QOL assessment was performed utilizing The Diabetes Treatment Satisfaction Questionnaires (DTSQ) for teens and for parents, separately [14]. The teens DTSQ contained 12 items scores on six-point scales, of which 9 were summed, the parents DTSQ contained 14 items, of which 9 were summed. Maximal grade was 42.
Skin reactions differences | 2 years from patient first enrollment
  skin assessment at the pump insertion site (itching and redness).
Discontinuation rate differences | 2 years from patient first enrollment
  Comparison between constant pump users and those who discontinued

SECONDARY OUTCOMES:
Glycemic control and metabolic parameters differences: Insulin TDD | 2 years from patient first enrollment
  The difference in glycemic control parameters and metabolic parameters after 3, 6 and 12 months of follow up, between the pumps devices. Insulin TDD, as reported by pump printout data
Glycemic control and metabolic parameters differences: HbA1c% | 2 years from patient first enrollment
  The difference in HbA1c% as measured by each center ll local lab.
Glycemic control and metabolic parameters differences:Glucose Mean & SD | 2 years from patient first enrollment
  Glucose Mean & SD as recorded by SMBG
Glycemic control and metabolic parameters differences:Number of SMBG per day | 2 years from patient first enrollment
  Data derived from data recorded by SMBG
Glycemic control and metabolic parameters differences:BMI SDS | 2 years from patient first enrollment
  according to Center for Disease Control (CDC) growth charts scale

IPD SHARING:
Plan to Share IPD: Undecided